CLINICAL TRIAL: NCT00441012
Title: A Study in Healthy Infants of the Safety, Tolerability, and Immunogenicity of Haemophilus Influenzae, Type b/Hepatitis B Vaccine Manufactured With a Modified Process
Brief Title: Study of Modified Process Hib/Hep B Vaccine in Infants (V121-019)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V121-019; 2007_513
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2009-07-10 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Haemophilus Influenzae Type B; Hepatitis B
Keywords: Haemophilus Influenza, type b and Hepatitis B
MeSH Terms: conditions — Haemophilus Infections; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Modified process Hib/Hep B vaccine
  Interventions: Biological: Comparator: Modified Process Vaccine
- 2 (Active Comparator): COMVAX™
  Interventions: Biological: Comparator: COMVAX™

INTERVENTIONS:
Biological: Comparator: Modified Process Vaccine — Modified process vaccine HBsAg 5 ug/0.5 mL and PRP [OMPC] 7.5 ug/0.5 mL in a 3-dose regimen at 2, 4 & 12 months of age. Duration of treatment is 11 months.
  Arms: 1
Biological: Comparator: COMVAX™ — COMVAX™ HBsAg 5 ug/0.5 mL and PRP [OMPC] 7.5 ug/0.5 mL in a 3-dose regimen at 2, 4, and 12 months of age. Duration of treatment is 11 months.
  Arms: 2

SUMMARY:
To determine if there is an improvement in the immune response to HBsAg (hepatitis B virus) in healthy infants using a modified process in a combination Haemophilus Influenzae, type b/Hepatitis B vaccine and a currently licensed Haemophilus Influenzae, type b/Hepatitis B vaccine

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month-old full term infants born to non-HBs Ag (hepatitis B virus) carrier mothers

Exclusion Criteria:

* Birth mother known to be a carrier of hepatitis B virus (HBsAg+) or known carriers ever living in close contact with the subject
* History of previous hepatitis B infection; history of vaccination with any hepatitis B vaccine
* Recent (<72 hours) history of febrile illness (rectal temperature >=38.1°C/>=100.5°F)
* Known or suspected hypersensitivity to any component of RECOMBIVAXHB™ or COMVAX™ (e.g., aluminum, yeast)
* Recent administration (w/i 3 months prior to study start) of hepatitis B immune globulin (HBIg), serum immune globulin, or any other blood-derived product
* Receipt of investigational drugs or investigational vaccines within 3 months prior to study start or if planned within the study period;
* Known or suspected impairment of immunologic function or recent use (within 3 months prior to study start) of immunomodulatory medications (does not include topical and inhaled steroids);
* Any condition that, in the opinion of the investigator, might interfere with the evaluation of study objectives; or inability to comply with the study schedule and/or inability to attend all required study visits

Ages: 40 Days to 80 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 546 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lee AW, Vesikari T, Gilbert CL, Klopfer SO, Schodel FP, Bhuyan PK. Immunogenicity and safety of a Haemophilus influenzae B (Hib)-hepatitis B vaccine with a modified process hepatitis B component administered with concomitant pneumococcal conjugate vaccine to infants. Vaccine. 2011 Oct 19;29(45):7942-8. doi: 10.1016/j.vaccine.2011.08.071. Epub 2011 Aug 27. PMID 21875633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 06-Dec-2006 (First Participant Enrolled in Study) to 03-Jun-2008 (Last Participant had their Last Visit).
  This study was conducted at 27 sites: 17 in Canada (16 of which were active sites) and 10 in Finland.
Pre-assignment Details: Participants excluded for history of or prior vaccination for hepatitis B (Hep B) or Haemophilus influenzae Type B (Hib) disease and for administration of blood products. Participants also excluded if mother received Hep B, Hib vaccine, or blood products 6 months prior to participant birth.
Groups:
- Modified Process Vaccine: Modified Process Vaccine (0, 2, and 10 months), 5/7.5 µg (micrograms)
- COMVAX™: COMVAX™ (0, 2, and 10 months), 5/7.5 µg (micrograms)
Period: Overall Study
Arm/Group | Modified Process Vaccine | COMVAX™
Started | 270 | 276
Vaccination Visit 1 | 269 (1 participant was randomized but not vaccinated in the Modified Process Vaccine group) | 276 (3 participants were vaccinated but were never randomized in the COMVAX™ group)
Vaccination Visit 2 | 267 | 272
Vaccination Visit 3 | 265 | 269
Completed | 252 | 263
Not Completed | 18 | 13
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 10 | 9
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Subject Randomized but Not Vaccinated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Modified Process Vaccine: Modified Process Vaccine (0, 2, and 10 months), 5/7.5 µg (micrograms)
  1 participant randomized but not vaccinated in the Modified Process Vaccine group; overall N is 269, not 270.
- COMVAX™: COMVAX™ (0, 2, and 10 months), 5/7.5 µg (micrograms)
  3 participants in the COMVAX™ group vaccinated but not randomized; overall N is 276, not 273 - due to issues randomizing via IVRS, in violation, all 3 participants were vaccinated as randomly assigned by the Investigator.
- Total: Total of all reporting groups
Arm/Group | Modified Process Vaccine | COMVAX™ | Total
Number analyzed (Participants) | 269 | 276 | 545
Age, Continuous [Mean (Standard Deviation); unit: Days] | 67.7 (8.9) | 68.3 (8.5) | 68.0 (8.7)
Age, Continuous [Mean (Full Range); unit: Days] | 67.7 [41 to 82] | 68.3 [40 to 83] | 68.0 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 142 | 271
  Male | 140 | 134 | 274

OUTCOME MEASURES:

1. Primary Outcome: The Number of Anti-HBs Seroprotected Participants 1 Month After the Third Dose.
Description: The number of participants as measured by the seroprotection rate (anti-hepatitis B surface antibodies greater than or equal to 10 mIU/mL). Anti-HBs (Antibodies against hepatitis B surface antigen) titers were measured from blood samples taken at Month 11 (1 month after the third dose)
Time Frame: 11 months (1 month after the third dose)
Population: Per-Protocol Population: The Per-Protocol Population is defined as the participants that were able to complete the study as defined by the protocol.
Measure: Number; unit: Participants
Arm/Group | Modified Process Vaccine | COMVAX™
Number analyzed (Participants) | 230 | 228
Participants | 230 | 226
Statistical Analysis 1: Comparison: Modified Process Vaccine; The purpose of the primary analysis is to demonstrate that there is an adequate seroprotection rate (percentage of participants with anti-HBs >=10mIU/mL) in each group at 1 month after the third dose. An adequate response requires the lower bound of the two-sided 95% confidence interval for the seroprotection rate to exceed 90%; Test type: Superiority or Other; Percentage of Seroprotected Participants = 100, 95% CI [98.7 to 100.0] — Exact binomial confidence interval
Statistical Analysis 2: Comparison: COMVAX™; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percentage of Seroprotected Participants = 99.1, 95% CI [69.9 to 99.9] — Exact binomial confidence interval

2. Primary Outcome: The Anti-HBs GMT (Geometric Mean Titer) 1 Month After the Third Dose.
Description: Geometric Mean Titer (GMT) - This is an Antibody titer that is measured using a laboratory test to detect the presence and amount of antibodies in a person's blood. Anti-HBs (Antibodies against hepatitis B surface antigen) and Geometric Mean Titers were measured from blood samples taken at Month 11 (1 month after the third dose).
Time Frame: 11 months (1 month after the third dose)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Modified Process Vaccine | COMVAX™
Number analyzed (Participants) | 230 | 228
mIU/mL | 4204.4 [3411.2 to 5182.0] | 1683.4 [1350.4 to 2098.6]
Statistical Analysis 1: Comparison: Modified Process Vaccine vs COMVAX™; Test type: Non-Inferiority or Equivalence — The Modified Process Vaccine is non-inferior to COMVAX with respect to anti-HBs GMT. The non-inferiority criterion requires that the lower bound of the two-sided 95% confidence interval on the ratio of the Month 11 GMTs [GMT modified process vaccine/GMT COMVAX™] is >0.67; Geometric Mean Titer Ratio = 2.5, 95% CI [1.9 to 3.3]

3. Secondary Outcome: The Total Number of Participants With Serious Vaccine-Related Clinical Adverse Experiences
Description: Participants with adverse experiences considered possibly, probably, or definitely related to study vaccines and considered serious (death, persistent disability, life threatening, hospitalization, birth defects, cancer, or overdose)
Time Frame: 0-11 months (recorded from first dose until the participant completes or discontinues)
Population: Safety Analysis Set: The Safety Analysis Set is defined as all participants who receive at least one injection of vaccine and who had a safety follow-up.
Measure: Number; unit: Participants
Arm/Group | Modified Process Vaccine | COMVAX™
Number analyzed (Participants) | 269 | 273
Participants | 0 | 0

4. Secondary Outcome: The Number of Anti-PRP Seroprotected Participants 1 Month After the Third Dose.
Description: The number of participants as measured by the seroprotection rate (anti-polyribosylribitol phosphate antibodies greater than 1 µg/mL). Anti-PRP (Antibodies against polyribosylribitol phosphate) titers were measured from blood samples taken at Month 11 (1 month after
  the third dose)
Time Frame: 11 months (1 month after the third dose)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Modified Process Vaccine | COMVAX™
Number analyzed (Participants) | 230 | 228
Participants | 216 | 210
Statistical Analysis 1: Comparison: Modified Process Vaccine; Test type: Superiority or Other; Percentage of Seroprotected Participants = 93.9, 95% CI [90.0 to 96.6] — Exact binomial confidence interval
Statistical Analysis 2: Comparison: COMVAX™; No hypothesis is being tested. The purpose of the secondary analysis is to estimate the seroprotection rate (percentage of participants with anti-PRP > 1µg/mL) in each group at 1 month after the third dose; Test type: Superiority or Other; Percentage of Seroprotected Participants = 92.1, 95% CI [87.8 to 95.3] — Exact binomial confidence interval

5. Secondary Outcome: The Anti-PRP GMT (Geometric Mean Titer) 1 Month After the Third Dose.
Description: Geometric Mean Titer (GMT) - This is an Antibody titer that is measured using a laboratory test to detect the presence and amount of antibodies in a person's blood. Anti-PRP (Antibodies against polyribosylribitol phosphate) titers were measured from blood samples taken at Month 11 (1 month after the third dose)
Time Frame: 11 months (1 month after the third dose)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | Modified Process Vaccine | COMVAX™
Number analyzed (Participants) | 230 | 228
µg /mL | 7.1 [6.0 to 8.4] | 8.0 [6.7 to 9.6]

ADVERSE EVENTS:
Arm/Group | Modified Process Vaccine | COMVAX™
Serious Adverse Events (participants affected / at risk) | 0 | 3
Other Adverse Events (participants affected / at risk) | 259 | 264
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Modified Process Vaccine | COMVAX™
Medication error (Injury, poisoning and procedural complications) | 0/269 | 1/273
Gastroenteritis (Infections and infestations) | 0/269 | 1/273
Gastroenteritis rotavirus (Infections and infestations) | 0/269 | 1/273
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Modified Process Vaccine | COMVAX™
Conjunctivitis (Eye disorders) | 6/269 | 8/273
Abdominal pain upper (Gastrointestinal disorders) | 6/269 | 6/273
Constipation (Gastrointestinal disorders) | 4/269 | 6/273
Diarrhea (Gastrointestinal disorders) | 24/269 | 26/273
Flatulence (Gastrointestinal disorders) | 8/269 | 14/273
Regurgitation (Gastrointestinal disorders) | 6/269 | 11/273
Teething (Gastrointestinal disorders) | 10/269 | 17/273
Vomiting (Gastrointestinal disorders) | 10/269 | 15/273
Fatigue (General disorders) | 19/269 | 15/273
Irritability (General disorders) | 117/269 | 131/273
Pyrexia (General disorders) | 162/269 | 167/273
Ear infection (Infections and infestations) | 5/269 | 3/273
Exanthema subitum (Infections and infestations) | 3/269 | 0/273
Gastroenteritis (Infections and infestations) | 3/269 | 3/273
Influenza (Infections and infestations) | 8/269 | 9/273
Laryngitis (Infections and infestations) | 0/269 | 4/273
Nasopharyngitis (Infections and infestations) | 8/269 | 11/273
Otitis media (Infections and infestations) | 12/269 | 12/273
Respiratory tract infection (Infections and infestations) | 3/269 | 2/273
Rhinitis (Infections and infestations) | 25/269 | 31/273
Upper respiratory tract infection (Infections and infestations) | 16/269 | 13/273
Body temperature increased (General disorders) | 6/269 | 8/273
Anorexia (Metabolism and nutrition disorders) | 14/269 | 10/273
Poor quality sleep (Nervous system disorders) | 4/269 | 3/273
Somnolence (Nervous system disorders) | 27/269 | 31/273
Crying (Psychiatric disorders) | 58/269 | 63/273
Insomnia (Psychiatric disorders) | 6/269 | 4/273
Restlessness (Psychiatric disorders) | 4/269 | 15/273
Cough (Respiratory, thoracic and mediastinal disorders) | 9/269 | 21/273
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6/269 | 8/273
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5/269 | 4/273
Eczema (Skin and subcutaneous tissue disorders) | 3/269 | 2/273
Erythema (Skin and subcutaneous tissue disorders) | 1/269 | 4/273
Rash (Skin and subcutaneous tissue disorders) | 14/269 | 10/273
Urticaria (Skin and subcutaneous tissue disorders) | 3/269 | 1/273
Injection site bruising (General disorders) | 9/269 | 9/273
Injection site erythema (General disorders) | 174/269 | 179/273
Injection site hematoma (General disorders) | 3/269 | 1/273
Injection site induration (General disorders) | 33/269 | 31/273
Injection site nodule (General disorders) | 6/269 | 6/273
Injection site pain (General disorders) | 195/269 | 213/273
Injection site swelling (General disorders) | 164/269 | 146/273

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.